CLINICAL TRIAL: NCT02449343
Title: A Registered Randomized, Double-Blind, Placebo-Controlled (2:1), Multi-Centered Clinical Trial of Anlotinib as a Treatment for Soft Tissue Sarcoma
Brief Title: Study of Anlotinib in Patients With Soft Tissue Sarcoma（STS）(ALTER0203)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-02-IIB
Record Dates: First submitted 2015-05-17; First posted 2015-05-20 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd
  Arms: Anlotinib
Drug: Placebo — Placebo p.o. qd
  Arms: Placebo

SUMMARY:
Compare the effects and safety of Anlotinib with placebo in patients with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Histological documentation of Soft Tissue Sarcoma,including Synovial sarcoma、Leiomyosarcoma、Alveolar soft part sarcoma、Undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma、Adipocytic Tumors、Fibrosarcoma、Clear cell sarcoma、Epithelioid sarcoma，With measurable disease.
* Within the past 6 months, using at least one failure of chemotherapy regimens (including anthracycline-based) in treating patients(except alveolar soft part sarcoma)
* 18-70years,ECOG PS:0-1,Life expectancy of more than 3 months
* Main organs function is normal
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it

Exclusion Criteria:

* Prior treatment with Anlotinib
* With pleural effusion or ascites, cause respiratory syndrome
* Accepted the vascular endothelial growth inhibitor class targeted drug treatment of patients
* Plan to take systemic anti-tumor therapy within 4 weeks before grouping or during the medicine-taking period of this research, including Cytotoxic Therapy, Signal Transduction Inhibitor, and Immunotherapy (or who use Mitomycin C within 6 weeks before taking the treatment with experimental drug); The patients who have already taken Extended Field Radiotherapy (EF-RT) within 4 weeks before grouping or Limited Field Radiotherapy with proposed assessment of nidus within 2 weeks before grouping
* Symptoms of brain metastases cannot be controlled and treated within less than 2 months
* With severe and failed to controlled diseases
* Occurred venous thromboembolic events within 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | up to 24 months

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months
Objective Response Rate (ORR) | up to 24 months
Disease Control Rate (DCR) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - The 1st Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Meidical University, Fuzhou, Fujian
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen university, Guangzhou, Guangdong
  - Guangxi medical university affiliated tumor hospital, Nanning, Guangxi
  - The Third Hospital of hebei Medical University, Shijiazhuang, Hebei
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - Henan Province Tumor Hospital, Luoyan, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xian Jiaotong University, Xian, Shanxi
  - West China Hospital , Sichuan University, Chengdu, Sichuan
  - Tianjin Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality